CLINICAL TRIAL: NCT02498444
Title: Perioperative Treprostinil in Pediatric Patients Undergoing the Fontan Operation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim futility analysis
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jeffrey A. Feinstein, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 33852
Record Dates: First submitted 2015-07-13; First posted 2015-07-15 (Estimated); Results first posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Single Ventricle
Keywords: Fontan; Treprostinil; Remodulin; Single ventricle
MeSH Terms: conditions — Univentricular Heart | interventions — treprostinil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treprostinil (Experimental): The subcutaneous continuous treprostinil infusion will start at a dose of 2 ng/kg/min. The dose will be increased over the first 24 hours to goal 10 ng/kg/min through day five. On postoperative day six, the dose will be decreased by 2 ng/kg/min every 8 hours with plans for discontinuation on postoperative day seven.
  Interventions: Drug: Treprostinil
- Saline (Placebo Comparator): Saline administration via subcutaneous infusion
  Interventions: Drug: Treprostinil

INTERVENTIONS:
Drug: Treprostinil — Administration of drug (treprostinil) vs placebo (saline) in the post-operative period
  Other Names: Remodulin

SUMMARY:
The purpose of this study is to test the efficacy of treprostinil (TRE) in the perioperative non-fenestrated, extracardiac Fontan patients in order to reduce duration of chest tube drainage (in days).

The Fontan operation is performed for patients with single ventricle physiology as the final palliation to create a series circulation, with passive systemic venous return to the pulmonary arteries and the single ventricle solely providing systemic output.

Patients undergoing extracardiac Fontan tend to have elevation of Fontan pressures immediately following the operation with inflammation from surgery requiring additional fluid administration to maintain blood pressure. Increased Fontan pressures and fluid overload lead to prolonged chest tube drainage.

The hypothesis is that treprostinil, a prostacyclin drug that dilates the pulmonary arteries, will improve immediate postoperative Fontan pressures. Treprostinil is not FDA approved for this use. Anecdotally and in a small case series, prostacyclin therapy has been shown to assist in transitioning patients off nitric oxide. The investigators believe that this improvement in hemodynamics will decrease duration of chest tube drainage resulting in a shorter length of hospital stay.

DETAILED DESCRIPTION:
In order to understand the effect of treprostinil on Fontan patients, this study has two parts:

1. reactivity testing with inhaled treprostinil in the cardiac catheterization lab for pre-Fontan patients undergoing routine catheterization in anticipation of the Fontan operation;
2. perioperative use of subcutaneous treprostinil starting immediately pre-op until postoperative day #7 to improve immediate postoperative hemodynamics and ultimately reduce overall length of hospital stay.

The investigators hope to learn how pulmonary vasodilator therapy affects and/or improves post- operative hemodynamics following the Fontan operation. This knowledge would be very important in the care of single ventricle patients following the Fontan operation if there is improvement of immediate outcomes and reduction of hospital length of stay. On a broader scale, if the use of treprostinil in perioperative Fontan patients can achieve the same results other centers achieve with the use of a fenestration this may have wide scale implications in the nationwide treatment of Fontan patients.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patient undergoing Fontan operation and/or pre-Fontan cardiac catheterization at Lucile Packard Children's Hospital (LPCH)

Exclusion Criteria:

* Platelet count < 50K (treprostinil can act as a platelet inhibitor and this may place patient at additional risk of bleeding if already thrombocytopenic)
* Dermatologic condition that renders the patient unable to tolerate a subcutaneous infusion (can still take part in inhaled vasodilator testing during cardiac catheterization)
* Currently receiving any vasodilator therapy specifically for the purpose of pulmonary vasodilation (phosphodiesterase type 5 inhibitor, endothelia receptor antagonist and/or prostacyclin).

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Feinstein, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Handler SS, Ogawa MT, Hopper RK, Sakarovitch C, Feinstein JA. Subcutaneous treprostinil in pediatric patients with failing single-ventricle physiology. J Heart Lung Transplant. 2017 Sep 14:S1053-2498(17)31993-9. doi: 10.1016/j.healun.2017.09.008. Online ahead of print. No abstract available. PMID 29126699

RESULTS

PARTICIPANT FLOW:
Groups:
- Treprostinil: Subcutaneous continuous treprostinil infusion starting at 2 ng/kg/min, increased over the first 24 hours to goal 10 ng/kg/min through day five, then decreased by 2 ng/kg/min every 8 hours starting on postoperative day six with plans for discontinuation on postoperative day seven.
Period: Overall Study
Arm/Group | Treprostinil | Saline
Started | 16 | 18
Completed | 12 | 18
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treprostinil | Saline | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 18 | 34
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 4.09 [3.35 to 4.82] | 4.51 [3.75 to 6.21] | 4.16 [3.50 to 4.96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 11 | 13 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 14
  Not Hispanic or Latino | 9 | 11 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 14 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 18 | 34
Ventricular morphology [Count of Participants; unit: Participants] — Description of the morphology of the functional systemic ventricle in this single ventricle congenital heart disease population
  Participants
    Left ventricle | 11 | 10 | 21
    Right ventricle | 5 | 8 | 13
Congenital Heart Disease [Count of Participants; unit: Participants] — Baseline congenital heart disease diagnosis
  Participants
    Hypoplastic left heart syndrome | 5 | 5 | 10
    Double inlet left ventricle | 5 | 4 | 9
    Tricuspid atresia | 3 | 3 | 6
    Double outlet right ventricle | 1 | 1 | 2
    Pulmonary atresia with intact ventricular septum | 2 | 2 | 4
    Atrioventricular septal defect | 0 | 2 | 2
    L-transposition of the great arteries + pulmonary atresia | 0 | 1 | 1
Baseline ventricular function [Count of Participants; unit: Participants] — Baseline ventricular function as measured by echocardiogram
  Participants
    Normal function | 15 | 15 | 30
    Mildly depressed function | 1 | 3 | 4
Systemic atrioventricular valve function [Count of Participants; unit: Participants] — Systemic atrioventricular valve function as measured by echocardiogram
  Participants
    No regurgitation | 1 | 3 | 4
    Trace regurgitation | 12 | 5 | 17
    Mild regurgitation | 2 | 6 | 8
    Mild-Moderate regurgitation | 1 | 2 | 3
    Moderate regurgitation | 0 | 2 | 2
Baseline Pulmonary Arterial Pressure [Median (Inter-Quartile Range); unit: mmHg] — Obtained on routine pre-operative cardiac catheterization.
  mmHg | 11.0 [9.75 to 12.0] | 9.0 [8.25 to 10.8] | 10.0 [9.0 to 12.0]
Baseline Atrial Pressure [Median (Inter-Quartile Range); unit: mmHg] — Obtained on routine pre-operative cardiac catheterization
  mmHg | 7.0 [5.0 to 8.0] | 5.0 [4.25 to 6.0] | 5.0 [5.0 to 7.25]
Baseline Transpulmonary Gradient [Median (Inter-Quartile Range); unit: mmHg] — Obtained on routine pre-operative cardiac catheterization
  mmHg | 4.0 [3.0 to 4.5] | 4.0 [4.0 to 5.0] | 4.0 [3.75 to 5.0]
Baseline Pulmonary Vascular Resistance [Median (Inter-Quartile Range); unit: indexed Wood units (WU*m^2)] — Obtained on routine pre-operative cardiac catheterization
  indexed Wood units (WU*m^2) | 1.12 [0.798 to 1.53] | 1.25 [1.06 to 1.56] | 1.2 [0.88 to 1.58]

OUTCOME MEASURES:

1. Primary Outcome: Chest Tube Duration
Description: This outcome measures the number of days that chest tubes were in place postoperatively.
Time Frame: 2-3 wks
Population: Intention to treat analysis based on study group assignment at randomization.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Treprostinil | Saline
Number analyzed (Participants) | 16 | 18
days | 8.0 [7.0 to 12.5] | 7.0 [5.0 to 8.0]
Statistical Analysis 1: Comparison: Treprostinil vs Saline; Test type: Other; p = 0.03, Poisson regression; Poisson regression model demonstrating associations between treatment groups and outcomes (chest tube duration in days and length of stay in days); Risk Ratio (RR) = 1.29, 95% CI 2-sided [1.02 to 1.64]

2. Secondary Outcome: Length of Hospital Stay
Description: This outcome measures the hospital length of stays in days.
Time Frame: 2-3 wks
Population: Intention to treat analysis based on group assignment at randomization
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Treprostinil | Saline
Number analyzed (Participants) | 16 | 18
days | 11.0 [9.5 to 14.5] | 9.0 [8.0 to 10.0]
Statistical Analysis 1: Comparison: Treprostinil vs Saline; Test type: Other; p = 0.0498, Poisson regression — Poisson regression model demonstrating associations between treatment groups and outcomes (chest tube duration in days and length of stay in days); Risk Ratio (RR) = 1.23, 95% CI 2-sided [1.00 to 1.51]

3. Secondary Outcome: Postoperative Fontan Pressure
Description: Patient hemodynamics as measured by invasive postoperative lines were recorded and compared between groups
Time Frame: postoperative hour 0, 12 and 24
Population: Participants with available data at the respective time points are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Treprostinil | Saline
Number analyzed (Participants) | 16 | 18
mmHg
  Fontan pressure- postoperative hour 0 | 13.0 [11.0 to 15.0] | 12.5 [11.0 to 13.25]
  Fontan pressure- postoperative hour 12: number analyzed (Participants) | 16 | 16
  Fontan pressure- postoperative hour 12 | 13.0 [12.25 to 15.0] | 10.5 [8.0 to 12.75]
  Fontan pressure- postoperative hour 24: number analyzed (Participants) | 13 | 13
  Fontan pressure- postoperative hour 24 | 13.0 [11.5 to 15.5] | 9.0 [8.0 to 15.5]
Statistical Analysis 1: Comparison: Treprostinil vs Saline; Between-group comparison at postoperative hour 0; Test type: Other; p = 0.05, Unadjusted repeated measure analysis
Statistical Analysis 2: Comparison: Treprostinil vs Saline; Between-group comparison at postoperative hour 12; Test type: Other; p < 0.01, Unadjusted repeated measure analysis
Statistical Analysis 3: Comparison: Treprostinil vs Saline; Between-group comparison at postoperative hour 24; Test type: Other; p = 0.14, Unadjusted repeated measure analysis

4. Secondary Outcome: Postoperative Atrial Pressure
Description: Patient hemodynamics as measured by invasive postoperative lines were recorded and compared between groups
Time Frame: postoperative hour 0, 12 and 24
Population: Participants with available data at the respective time points are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Treprostinil | Saline
Number analyzed (Participants) | 16 | 17
mmHg
  Postoperative hour 0: number analyzed (Participants) | 15 | 17
  Postoperative hour 0 | 7.0 [5.0 to 9.0] | 5.0 [4.0 to 7.0]
  Postoperative hour 12: number analyzed (Participants) | 16 | 16
  Postoperative hour 12 | 6.0 [5.0 to 8.75] | 6.0 [4.0 to 8.0]
  Postoperative hour 24: number analyzed (Participants) | 7 | 8
  Postoperative hour 24 | 6.0 [5.0 to 12.0] | 7.0 [4.25 to 10.75]
Statistical Analysis 1: Comparison: Treprostinil vs Saline; Between-group comparison at postoperative hour 0; Test type: Other; p = 0.23, Unadjusted repeated measure analysis
Statistical Analysis 2: Comparison: Treprostinil vs Saline; Between-group comparison at postoperative hour 12; Test type: Other; p = 0.27, Unadjusted repeated measure analysis
Statistical Analysis 3: Comparison: Treprostinil vs Saline; Between-group comparison at postoperative hour 24; Test type: Other; p = 0.65, Unadjusted repeated measure analysis

5. Secondary Outcome: Postoperative Transpulmonary Gradient
Description: Patient hemodynamics as measured by invasive postoperative lines were recorded and compared between groups. Transpulmonary pressure gradient is defined as the difference between mean pulmonary artery pressure and left atrial pressure (commonly estimated by a pulmonary artery wedge pressure).
Time Frame: postoperative hour 0, 12 and 24
Population: Participants with available data at the respective time points are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Treprostinil | Saline
Number analyzed (Participants) | 16 | 17
mmHg
  Postoperative hour 0: number analyzed (Participants) | 15 | 17
  Postoperative hour 0 | 7.0 [5.0 to 8.0] | 7.0 [5.0 to 7.5]
  Postoperative hour 12: number analyzed (Participants) | 16 | 16
  Postoperative hour 12 | 7.0 [5.0 to 9.75] | 4.0 [3.25 to 5.0]
  Postoperative hour 24: number analyzed (Participants) | 7 | 8
  Postoperative hour 24 | 6.0 [5.0 to 10.0] | 6.0 [4.0 to 7.0]
Statistical Analysis 1: Comparison: Treprostinil vs Saline; Between-group comparison at postoperative hour 0; Test type: Other; p = 0.37, Unadjusted repeated measure analysis
Statistical Analysis 2: Comparison: Treprostinil vs Saline; Between-group comparison at postoperative hour 12; Test type: Other; p < 0.01, Unadjusted repeated measure analysis
Statistical Analysis 3: Comparison: Treprostinil vs Saline; Between-group comparison at postoperative hour 24; Test type: Other; p = 0.30, Unadjusted repeated measure analysis

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during hospitalization, which was generally between 1-3 weeks.
Arm/Group | Treprostinil | Saline
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/18
Other Adverse Events (participants affected / at risk) | 7/16 | 0/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treprostinil (N=16) | Saline (N=18)
Site pain (General disorders) | 7 | 0 (0) — Pain related to subcutaneous catheter site

LIMITATIONS AND CAVEATS:
Early termination based on futility analysis performed prior to full study enrollment led to smaller number of subjects analyzed than initially outlined by power analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT02498444/Prot_SAP_000.pdf